CLINICAL TRIAL: NCT01471743
Title: The Effect of Pre-Operative Immunonutrition With "Impact Advanced Recovery (R)" on Patients Undergoing Major GI Cancer Surgery
Brief Title: GI Surgery Pre-Operative Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sherri L Lewis, Chief, Clinical Nutrition, James A. Haley Veterans Administration Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00002602
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Immunonutrition
Keywords: nutrition; surgery; immune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impact Advance Recovery (R) (Experimental): 3 supplements per day for 5 days pre-operatively
  Interventions: Dietary Supplement: Impact Advance Recovery (R)
- Standard Supplement (Active Comparator): 3 supplement per day for 5 days pre-operatively
  Interventions: Dietary Supplement: Ensure Plus (R)

INTERVENTIONS:
Dietary Supplement: Impact Advance Recovery (R)
  Arms: Impact Advance Recovery (R)
Dietary Supplement: Ensure Plus (R)
  Arms: Standard Supplement

SUMMARY:
Surgical patients are high risk for post operative infections. These post operative infections contribute to increased length of hospital stay, hospital costs and delay overall recovery time thus decreasing the quality of life. Studies have reported post operative complications ranging from 37% to 74%.1 The most costly complications include infectious complications after major Gastrointestinal (GI) surgery including wound infections, abdominal abscess, pneumonia, sepsis and anastomic leaks.2 Several studies have been conducted that show a significant reduction in infectious complications and average length of stay when treated with immunonutrition supplements.2-3 A review of similarly designed studies in a different patient population indicate that post-operative infections can be reduced by an average of 71% with immunonutrition.

This study seeks to investigate the effect of Impact Advanced Recovery ® in improving surgical outcomes in patients receiving major gastrointestinal surgeries compared to a standard supplement at James A. Haley Veterans' Hospital. Providing Impact Advanced Recovery ® may decrease post-operative infectious complications, length of stay, and recovery time.

Hypothesis

1. In patients receiving elective gastrointestinal surgery (esophageal, gastric, pancreatic or colon resections) there will be a significant decrease of at least 60% in post-operative infections as listed below for patients who consume 15 servings of Impact Advanced Recovery® pre-operatively compared to patients who consume 15 servings of a standard supplement.

   Complications to be considered: anastomatic leak, post-op wound development, post-op abdominal abscess, sepsis, pneumonia, post-op ileus, intestinal fistula, obstruction, urinary tract infections, peritonitis or bowel necrosis.
2. In patients receiving elective gastrointestinal surgery (esophageal, gastric, pancreatic or colon resections) there will be a significant decrease in hospital and NPO days for patients who consume 15 servings of Impact Advanced Recovery ® pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented neoplasm of the gastrointestinal tract.
* Planned major elective surgery including esophageal, gastric, pancreatic or colon resections.

Exclusion Criteria:

* Critically ill patients defined as any patient admitted to the intensive care unit (ICU) prior to elective surgery.
* Current use of steroids or other immunosuppressive medications.
* History of hospitalization for pulmonary, cardiac or renal disease in the 6 months prior to elective surgery.
* Patients who exhibit signs and symptoms of infection or sepsis including: elevated WBC above 10,000 cells/ml; temperature > 37.7 C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with post-op Infections | within 30 days post-operatively
  Determine the effectiveness of pre-operative supplementation with Impact Advanced Recovery ® on reducing the risk of developing complications during the 30 day post-operative period with decreased length of hospital stay, and time to resume an oral diet.

CONTACTS AND LOCATIONS:
Locations (1):
- James A. Haley VA Hospital, Tampa, Florida, United States